CLINICAL TRIAL: NCT07225244
Title: Comparative Outcomes of Four Versus Two Balloon Inflation Points in Dacryoplasty for Primary Acquired Nasolacrimal Duct Obstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202509023RIND
Record Dates: First submitted 2025-11-03; First posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Primary Acquired Nasolacrimal Duct Obstruction
Keywords: balloon dacryoplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 4-point group (Experimental): Balloon dacryoplasty with LacriCATH® at 4 different points in the nasolacrimal duct
  Interventions: Device: 4 point balloon dacryoplasty with LacriCATH®
- 2-point group (Active Comparator): Balloon dacryoplasty with LacriCATH® at 2 different points in the nasolacrimal duct
  Interventions: Device: 2 point balloon dacryoplasty with LacriCATH®

INTERVENTIONS:
Device: 2 point balloon dacryoplasty with LacriCATH® — Balloon dacryoplasty with LacriCATH® (QUEST Medical Inc., Allen, TX, USA, 3 mm balloon diameter, 15 mm in length). The balloon will be inflated to 8 bars of pressure for 90 seconds, deflated, and re-inflated to 8 bars of pressure for an additional 90 seconds at two different points.
  Arms: 2-point group
Device: 4 point balloon dacryoplasty with LacriCATH® — Balloon dacryoplasty with LacriCATH® (QUEST Medical Inc., Allen, TX, USA, 3 mm balloon diameter, 15 mm in length). The balloon will be inflated to 8 bars of pressure for 90 seconds and deflated at four different points.
  Arms: 4-point group

SUMMARY:
Primary acquired nasolacrimal duct obstruction

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary acquired nasolacrimal duct obstruction (PANDO)

Exclusion Criteria:

* Patients who are pregnant, with previous lacrimal procedure, upper lacrimal drainage obstruction, punctal stenosis, active dacryocystitis, dacryolithiasis, traumatic obstruction or lacrimal mass

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Munk's scale for epiphora grading | From enrollment to 6 months after intervention
  The frequency of epiphora will be evaluated at each follow-up visit using the Munk's scale, in which patients rate the frequency of tearing on a standardized 0-5 scale based on daily symptoms (as below).
  Grade 0: no epiphora Grade 1: epiphora requiring dabbing less than twice a day Grade 2: epiphora requiring dabbing 2-4 times a day Grade 3: epiphora requiring dabbing 5-10 times a day Grade 4: epiphora requiring dabbing more than 10 times a day Grade 5: constant epiphora
  The higher the grade, the worse the condition.

SECONDARY OUTCOMES:
Tear meniscus height | For enrollment to 6 months after intervention
  Tear meniscus height (TMH) will be objectively measured using the OCULUS Keratograph 5M, a noninvasive ocular surface analyzer. The measurement will be recorded in millimeters (mm) at each visit to assess tear volume and lacrimal drainage function.
Patency of the nasolacrimal system assessed by probing and irrigation of the nasolacrimal duct | For enrollment to 6 months after intervention
  Patency of the nasolacrimal drainage system will be evaluated by performing probing and irrigation of the nasolacrimal duct under topical anesthesia. The outcome will be categorized as patent, partially obstructed, or completely obstructed based on the ease of probe passage and saline flow into the nasal cavity.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsuan Wei, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No